Nothing herein is to be disclosed in any way without the prior express written permission of W. L. Gore & Associates, Inc.

Assessment of the GORE® EXCLUDER® Conformable AAA Endoprosthesis in the Treatment of Abdominal Aortic Aneurysms

Protocol number: AAA 13-03

07September2022

W. L. Gore & Associates, Inc. Medical Products Division

## **PROTOCOL SUMMARY**

| Study Title | Assessment of the GORE® EXCLUDER® Conformable AAA Endoprosthesis (CEXC Device) in the Treatment of Abdominal Aortic Aneurysms |
|---|---|
| Protocol Number | AAA 13-03 |
| IDE or PMA Number | IDE # G150057 |
| Sponsor | W. L. Gore & Associates, Inc. |
| | Telephone: 800-437-8181 |
| Study Design | Prospective, nonrandomized, multicenter, study with two parallel substudies: |
| | Short Neck Substudy: Subjects with abdominal aortic aneurysms having aortic neck angulation ≤ 60° and infrarenal aortic neck length ≥ 10 mm |
| | High Neck Angulation Substudy: Subjects with abdominal aortic aneurysms having aortic neck angulation > 60 °and ≤ 90° and infrarenal aortic neck length ≥ 10 mm |
| Study Objective | Assess the safety and effectiveness of the CEXC Device for the treatment of infrarenal AAA |
| Primary Safety<br>Endpoint (Both<br>Substudies) | <ul> <li>Composite of any of the following events through 30 days post-treatment:</li> <li>Death</li> <li>Stroke</li> <li>Myocardial Infarction</li> <li>Bowel Ischemia</li> <li>Paraplegia</li> <li>Respiratory Failure</li> <li>Renal Failure</li> <li>Blood Loss &gt; 1000 mL</li> <li>Thromboembolic Events (including limb occlusion and distal embolic events)</li> </ul> |

| Primary Safety<br>Endpoint Hypothesis<br>(Both Substudies) | Percentage of subjects free from safety events as adjudicated by the Clinical Events Committee (CEC) at 30 days will be > 79% |
|---|---|
| Primary Effectiveness<br>Endpoint (Both<br>Substudies) | Treatment success, defined as technical success (defined as successful access and deployment of all required CEXC Device components) and freedom from the following events: |
| | <ul> <li>Type I endoleak</li> <li>Type III endoleak</li> <li>Migration (10 mm or more)</li> <li>AAA enlargement ≥ 5 mm with or without intervention</li> <li>AAA rupture</li> <li>Conversion to open repair</li> </ul> |
| Primary Effectiveness<br>Endpoint Hypothesis<br>(Both Substudies) | The percentage of subjects with treatment success at one year will be > 80% |
| Subject Population | Subjects with infrarenal abdominal aortic aneurysm (AAA) |
| | Initial Cohort: A total of 175 subjects: |
| Number of Subjects | 80 Short Neck Substudy, 95 High Neck Angulation Substudy |
| · | Continued Enrollment Cohort (optional): Up to 15 High Neck Angulation Subjects. |
| Number of Sites | A maximum of 56 sites located in the U.S. |
| | The Sponsor shall maintain an updated list of principal investigators, investigational sites, and institutions. This list shall be kept separately from this Protocol. |
| Expected Time to | Subject accrual – 2 years |
| Complete Enrollment | Follow-up – 5 years from last subject enrollment |
| | Total investigation duration – 10 years |
| | (including site initiation and closing period) |
| Expected Time of each Study Subject to Complete the Study | Total of 60 months for each subject to complete the study |
| Pre-Treatment<br>Evaluation | <ul> <li>Physical exam / medical history within 30 days of procedure</li> <li>Serum creatinine concentration</li> <li>Contrast enhanced spiral CT of the abdomen and pelvis ≤ 90 days from procedure</li> </ul> |
| Follow-Up Evaluations | Follow-up conducted at one, six, and twelve months post-treatment and annually thereafter for five years to consist of: • Physical examination • Contrast enhanced CT scan |
| | Non-contrast CT scan (1 month only) |

| Cinnificant Includes | |
|---|---|
| Significant Inclusion<br>Criteria | <ul> <li>AAA meeting any of the following criteria:</li> <li>Maximum diameter ≥ 50 mm</li> <li>Rapid growth (&gt; 5 mm in a 6 month period)</li> <li>Non-ruptured AAA presenting with clinical symptoms</li> <li>Adequate anatomy to receive the CEXC Device, including:</li> <li>Adequate iliac / femoral access</li> <li>Infrarenal aortic neck diameter 16-32 mm</li> <li>Infrarenal aortic neck length ≥ 10 mm</li> <li>Aortic neck angle ≤ 90°</li> <li>Distal iliac artery seal zone ≥ 10 mm</li> <li>Iliac artery diameter 8-25 mm</li> <li>An Informed Consent Form (ICF) signed by subject</li> <li>Male or infertile female*</li> <li>Able to comply with Protocol requirements including following-up</li> <li>Life expectancy &gt; 2 years</li> <li>Age ≥ 21 years</li> <li>* Infertile female – condition which prevents pregnancy, e.g., hysterectomy, tubal ligation or postmenopausal for greater than 1 year</li> <li>Subjects will be allocated to the appropriate substudy based on the aortic neck angle measurement recorded during screening.</li> </ul> |
| Significant Exclusion<br>Criteria | <ul> <li>Mycotic or ruptured aneurysm</li> <li>Known concomitant thoracic aortic aneurysm which requires surgical intervention</li> <li>Renal insufficiency defined as creatinine &gt; 2.5 mg / dL or patient undergoing dialysis</li> <li>New York Heart Association (NYHA) class IV</li> <li>Aneurysmal, dissected, heavily calcified, or heavily thrombosed landing zone(s)</li> <li>Severely tortuous or stenotic iliac and / or femoral arteries</li> <li>Patient has body habitus or other medical condition which prevents adequate delineation of the aorta</li> <li>Participating in another investigational device or drug study within 1 year of treatment</li> </ul> |

| | <ul> <li>Systemic infection which may increase the risk of endovascular graft infection</li> <li>Known degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome</li> <li>Planned concomitant surgical procedure or major surgery within 30 days of treatment date</li> <li>Known history of drug abuse</li> <li>Known sensitivities or allergies to the device materials</li> </ul> |
|---|---|
| Total Expected Duration of the Study | Total investigation duration – 10 years (including site initiation and closing period) |
| Schedule of Events-<br>All Enrolled Subjects | Screening Pre-Treatment Treatment Discharge Follow-up (30 day, 6 and 12 month and annually through 5 years). |
| Data Monitoring<br>Committees | Clinical Events Committee (CEC) Data Safety Monitoring Board (DSMB) |